CLINICAL TRIAL: NCT03320057
Title: Alternative Provision of Medication Abortion Via Pharmacy Dispensing
Brief Title: Medication Abortion Via Pharmacy Dispensing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daniel Grossman (Other)
Collaborators: University of California, San Diego (Other); University of California, Davis (Other); University of Washington (Other); Kaiser Permanente (Other); Planned Parenthood of the Great Northwest and Hawaiian Islands (Other)
Responsible Party: Sponsor-Investigator, Daniel Grossman, Professor in Dept ObGyn and Director of Advancing New Standards in Reproductive Health, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: A128753
Record Dates: First submitted 2017-09-26; First posted 2017-10-25 (Actual); Results first posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Pregnancy Related; Abortion Early
Keywords: medication abortion; mifepristone
MeSH Terms: interventions — Mifepristone

STUDY DESIGN:
Intervention Model Description: Prospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Medication abortion patients (Experimental): Oral mifepristone 200 mg, followed by misoprostol 800 mcg administered buccally (at 24-48 hours following mifepristone) or vaginally (as soon as 6 hours following mifepristone)
  Interventions: Drug: Mifepristone
- Pharmacists (Other): Pharmacists providing services at one of the study pharmacies during the study
  Interventions: Other: Training on mifepristone dispensing

INTERVENTIONS:
Drug: Mifepristone — Patients will receive Mifeprex® (mifepristone) by pharmacy rather than standard care at clinic visit
  Arms: Medication abortion patients
Other: Training on mifepristone dispensing — Pharmacists were offered a training on medication abortion and mifepristone dispensing
  Arms: Pharmacists

SUMMARY:
This mixed-methods study follows a prospective cohort of patients receiving Mifeprex ® (mifepristone) for medication abortion dispensed by pharmacists after undergoing standard clinical evaluation. Women participating in this study will obtain mifepristone and misoprostol from the pharmacy instead of in the clinic. To assess feasibility, acceptability, and effectiveness of pharmacy dispensing of mifepristone, the study will survey patients, evaluate their clinical outcomes from electronic health records, and survey and interview pharmacists at study sites.

DETAILED DESCRIPTION:
Improving access to and efficiency of abortion provision is important for patients and providers. The Risk Evaluation and Mitigation Strategy (REMS) requires that Mifeprex ® ( mifepristone) be dispensed only from a doctor's office, clinic or hospital (not from a pharmacy by prescription) by a certified health care provider and the health care provider must obtained a signed Patient Agreement Form before dispensing mifepristone. Data are needed to investigate the feasibility, acceptability, and effectiveness of pharmacy dispensing of mifepristone. In order to address the study question, a mixed methods study design is appropriate. To assess feasibility, the study will collect data on pharmacists' satisfaction with dispensing mifepristone. To assess acceptability, qualitative data will be collected from pharmacists about their perspectives on dispensing Mifeprex before and after the study, as well as measure patient satisfaction through open-ended and close-ended survey questions. To assess effectiveness of the pharmacy dispensing model, the study will evaluate clinical outcomes from electronic health records. The proposed feasibility study would take place at sites in California and Washington states.

ELIGIBILITY:
Patient Inclusion Criteria:

* Women seeking medication abortion through 70 days gestation
* Eligible for Mifeprex® at a study clinical site
* English or Spanish speaking
* Willing and able to participate in the study, including willing to go to the study pharmacy to obtain mifepristone

Patient Exclusion Criteria:

* Not pregnant
* Not seeking medication abortion
* Under the age of 15
* Contraindications for medication abortion

  * All pharmacists providing services at one of the study pharmacies during the study are eligible for the pharmacist survey and interview.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Females seeking medication abortion
Enrollment: 326 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-07-04 (Actual); Study Completion 2020-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Grossman, MD, Principal Investigator — University of California, San Francisco
Locations (6):
- United States (6):
  - Obstetrics and Gynecology Family Planning Clinic at University of California Davis, Sacramento, California
  - Women's Health Services at University of California San Diego, San Diego, California
  - Kaiser Permanente Northern California, San Francisco, California
  - Mt. Zion Women's Options Clinic, University, San Francisco, California
  - University of Washington, Seattle, Washington
  - Planned Parenthood Great Northwest, Hawai'i, Alaska, Indiana, Kentucky, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaller S, Morris N, Biggs MA, Baba CF, Rafie S, Raine-Bennett TR, Creinin MD, Berry E, Micks EA, Meckstroth KR, Averbach S, Grossman D. Pharmacists' knowledge, perspectives, and experiences with mifepristone dispensing for medication abortion. J Am Pharm Assoc (2003). 2021 Nov-Dec;61(6):785-794.e1. doi: 10.1016/j.japh.2021.06.017. Epub 2021 Jun 18. PMID 34281806
- [Derived] Grossman D, Baba CF, Kaller S, Biggs MA, Raifman S, Gurazada T, Rafie S, Averbach S, Meckstroth KR, Micks EA, Berry E, Raine-Bennett TR, Creinin MD. Medication Abortion With Pharmacist Dispensing of Mifepristone. Obstet Gynecol. 2021 Apr 1;137(4):613-622. doi: 10.1097/AOG.0000000000004312. PMID 33706339

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient Recruitment: Study recruitment began in July 2018 and was halted before reaching our desired sample size in March 2020 owing to the coronavirus disease 2019 (COVID-19) pandemic, which limited the ability to have research staff in clinical facilities and lengthen patient visits for the purposes of research consent.
  Pharmacist Recruitment: We invited all pharmacists providing services at the study pharmacies to participate in the study and dispense mifepristone to study patients.
Pre-assignment Details: Research staff assessed 499 patients for eligibility, of whom 233 were ineligible (n=163) or declined to participate (n=70). We enrolled 266 patient participants, all of whom received the study medications from the pharmacy. We invited 72 pharmacists working at six study pharmacy sites to participate in the study, including training to dispense mifepristone and completion of the baseline survey.
Groups:
- Pharmacist Providing Services at One of the Study Pharmacies During the Study: All pharmacists providing services at one of the study pharmacies during the study were invited to participate in the training on dispensing mifepristone and surveys. Only trained pharmacists were eligible to participate in the endline survey.
Period: Overall Study
Arm/Group | Medication Abortion Patients | Pharmacist Providing Services at One of the Study Pharmacies During the Study
Started | 266 | 60 (Includes pharmacists at study pharmacies that consented to training on mifepristone dispensing.)
Patient's Clinical Outcome Information Obtained | 262 | 0 (Clinical outcome data were not collected for pharmacists - this milestone does not apply)
Received Pharmacist Training | 0 | 56
Pharmacists Completed Baseline Survey | 0 | 47
Completed | 260 | 43 (This includes pharmacists who completed the endline survey. Only trained pharmacists (n=56) were eligible.)
Not Completed | 6 | 17
Not completed — Lost to Follow-up | 4 | 17
Not completed — Did not take mifepristone or misoprostol | 2 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes patient study participants having medication abortion and receiving mifepristone at a study pharmacy. Pharmacist participants are not reported here as baseline demographics were not collected from them.
Arm/Group | Medication Abortion Patients
Number analyzed (Participants) | 260
Age, Continuous [Median (Full Range); unit: years] | 28 [16 to 44]
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical: 16-20 years | 22
  Age, Categorical: 21-24 years | 45
  Age, Categorical: 25-29 years | 78
  Age, Categorical: 30-34 years | 69
  Age, Categorical: 35-44 years | 46
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex/Gender Not Collected
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and ethnicity, Categorical: Non-Hispanic White | 99
  Race and ethnicity, Categorical: Non-Hispanic Black | 29
  Race and ethnicity, Categorical: Hispanic | 65
  Race and ethnicity, Categorical: Asian or Pacific Islander | 45
  Race and ethnicity, Categorical: Alaska Native or Native American | 2
  Race and ethnicity, Categorical: Other and mixed race and ethnicity | 19
  Race and ethnicity, Categorical: Missing | 1
Region of Enrollment [Number; unit: participants]
  United States | 260
Education, Categorical [Count of Participants; unit: Participants]
  High school or less | 39
  Some college or professional school | 93
  College degree | 90
  Advanced degree | 28
  Missing | 10
Relationship status, Categorical [Count of Participants; unit: Participants]
  Neither married nor in a relationship | 84
  Married | 54
  Committed relationship | 110
  Missing | 12
Parity [Count of Participants; unit: Participants]
  Nulliparous | 171
  Parous | 89
History of abortion, Categorical [Count of Participants; unit: Participants]
  None | 165
  Previous medication abortion | 48
  Previous procedural abortion only | 40
  Missing | 7
Gestational age at initial visit, Continuous [Median (Full Range); unit: days] | 46 [30 to 70]
Gestational age at initial visit, Categorical [Count of Participants; unit: Participants]
  49 days or less | 176
  50-56 days | 43
  57-63 days | 32
  64-70 days | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Pharmacists Who Objected to Participate in Dispensing Mifeprex
Description: Number of pharmacists who objected to participate in dispensing Mifeprex at least once during the study period. This includes pharmacists who declined participation in the study training on medication abortion due to discomfort as well as pharmacists who participated in the training but declined to dispense Mifeprex.
Time Frame: End of the study, month 24
Population: Pharmacists invited to participate in mifepristone dispensing
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacists
Number analyzed (Participants) | 72
Participants | 4

2. Primary Outcome: Number of Pharmacists Who Report Being Satisfied With Pharmacy Dispensing of Mifeprex
Description: Number of pharmacists who report being "somewhat satisfied" or "very satisfied" when asked "Overall, how satisfied are you with mifepristone dispensing at your pharmacy?" in endline survey
Time Frame: End of the study, month 24
Population: Pharmacists at study pharmacist who were trained to dispense mifepristone and completed an endline survey
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacists
Number analyzed (Participants) | 43
Participants | 36

3. Secondary Outcome: Number of Participants Who Report Being Satisfied With Obtaining Mifeprex in the Pharmacy
Description: Number of participants who report being "somewhat satisfied" or "very satisfied" when asked "Overall, how satisfied were you with your experience at the pharmacy when you got the abortion pill?"
Time Frame: Day 2 following initial medication abortion visit
Population: Patient participants who completed Day 2 survey following initial medication abortion visit
Measure: Count of Participants; unit: Participants
Arm/Group | Medication Abortion Patients
Number analyzed (Participants) | 252
Participants | 230

4. Secondary Outcome: Number of Participants With a Complete Abortion With Medication Alone and Who do Not Require a Surgical Procedure to Complete the Abortion
Description: Number of participants who report that their "abortion is now complete and they are no longer pregnant" and who did not "end up having a suction procedure (or vacuum aspiration or dilation and curettage procedure) to complete the abortion"
Time Frame: Up to 6 weeks after initial visit
Population: Patient participants with abortion outcome information
Measure: Count of Participants; unit: Participants
Arm/Group | Medication Abortion Patients
Number analyzed (Participants) | 260
Participants | 243

5. Secondary Outcome: Number of Participants With an Adverse Event
Description: Number of participants who had a medical problem that required them to go to the hospital, emergency department or a doctor's office (other than regularly scheduled follow-up visit) since receiving the abortion pill
Time Frame: Up to 6 weeks after initial visit
Population: Patients with follow-up data from clinical data or survey responses
Measure: Count of Participants; unit: Participants
Arm/Group | Medication Abortion Patients
Number analyzed (Participants) | 260
Participants | 4

6. Secondary Outcome: Difference in Pharmacists' Mean Knowledge Score Related to Medication Abortion
Description: Difference in pharmacists' mean knowledge score related to medication abortion. Knowledge scores were based on a set of 15 statements or questions related to medication abortion for which respondents selected answer(s) from multiple choice response options. Topics included medication abortion dosing regimen, biological processes during medication abortion, clinical outcomes, and federal and state policies relating to medication abortion. For pharmacists who had completed at least 50% of the items, we calculated their average number of correct responses among completed items, as a proportion of correct answers, ranging from 0-1, with 1 meaning 100% correct. All questions or statements included an "I don't know" response option, which we coded as incorrect. Higher scores mean a higher level of knowledge.
Time Frame: Before and after the intervention, approximately month 1 and month 18 of the study to assess differences in knowledge
Population: We compared knowledge scores for pharmacists at baseline and endline. We excluded from the baseline knowledge analyses four respondents who participated in the study training on medication abortion prior to taking the baseline survey and one person from the overall knowledge analyses because they only completed four items.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pharmacists
Number analyzed (Participants) | 53
score on a scale
  Baseline knowledge score: number analyzed (Participants) | 43
  Baseline knowledge score | 0.51 (0.21)
  Endline knowledge score: number analyzed (Participants) | 43
  Endline knowledge score | 0.64 (0.24)
Statistical Analysis 1: Comparison: Pharmacists; Medication abortion knowledge scores were based on a set of 15 items. We first assessed the internal consistency reliability of the 15 knowledge items and considered a Cronbach's alpha coefficient above .70 to be acceptable to examine the items as a combined score; Test type: Other — We conducted multivariable logistic regression analyses using Generalized Estimating Equation (GEE) models to assess whether study implementation was associated with pharmacists' overall medication abortion knowledge. Multivariable GEE analyses included time period (baseline and endline) as the primary independent variable, adjusted for gender and years of experience, and accounted for clustering by pharmacy site and individual pharmacist; p < 0.05, Regression, Linear; Beta Coefficient = 0.14, 95% CI 2-sided [0.11 to 0.17] — Coefficients in adjusted analyses examining overall medication abortion knowledge represent the difference in mean knowledge scores between baseline and endline

ADVERSE EVENTS:
Time Frame: Patients: Up to 6 weeks after initial visit Pharmacists: study duration including training, mifepristone dispensing, survey data collection (approximately 24 months)
Description: Patients: A medical problem that required patients to go to the hospital, emergency department or a doctor's office (other than regularly scheduled follow-up visit) since receiving the abortion pill.
  Pharmacists: Any untoward/unfavorable medical occurrence, including any abnormal sign, symptom, or disease, temporally associated with participation in training, mifepristone dispensing, or survey data collection, whether or not considered related to their participation in the research.
Groups:
- Pharmacists: Pharmacists providing services at one of the study pharmacies during the study and consenting to training
Arm/Group | Medication Abortion Patients | Pharmacists
All-Cause Mortality (participants affected / at risk) | 0/260 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/260 | 0/60
Other Adverse Events (participants affected / at risk) | 4/260 | 0/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medication Abortion Patients (N=260) | Pharmacists (N=60)
Dehydration (General disorders) | 1 (1) | 0
Heavy uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 — Uterine bleeding is a normal part of the medication abortion process, however, bleeding is reported here as an adverse event because it caused the participant to go to the emergency department
Pelvic Inflammatory Disease (Reproductive system and breast disorders) | 1 (1) | 0 — Diagnosis of pelvic inflammatory disease after aspiration for incomplete medication abortion
Swelling in cheeks (Skin and subcutaneous tissue disorders) | 1 (1) | 0 — Swelling in cheeks and transient pain in cheeks after taking misoprostol buccally, thought to be a possible allergic reaction

LIMITATIONS AND CAVEATS:
We aimed to recruit 300-350 patients for this study. We had to stop recruitment early because of the COVID-19 pandemic, reaching 89% of our planned minimum sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT03320057/Prot_006.pdf
  • Statistical Analysis Plan (2021-05-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT03320057/SAP_007.pdf